CLINICAL TRIAL: NCT00000939
Title: Phase II Randomized, Open-Label Study of Maintenance of HIV RNA Suppression After Switching to ddI/d4T/HU vs. ddI/d4T/EFV vs. Continuing the Pre-Entry Protease Inhibitor Regimen
Brief Title: A Study to Compare the Effectiveness of Different Anti-HIV Drug Regimens in Keeping Levels of HIV in the Blood as Low as Possible
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A5039; 10885 (Registry Identifier: DAIDS ES); ACTG A5039
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Hydroxyurea; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; efavirenz; Stavudine; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Efavirenz
Drug: Stavudine
Drug: Didanosine

SUMMARY:
This study will look at different anti-HIV drug regimens to see which works best to keep the level of HIV (viral load) in the blood as low as possible during maintenance therapy. You will be assigned randomly (like tossing a coin) to 1 of 3 groups:

Group 1: Didanosine plus stavudine plus hydroxyurea (ddI/d4T/HU). Group 2: Didanosine plus stavudine plus efavirenz (ddI/d4T/EFV). Group 3: This group of patients will remain on their current drug regimens. This study will last approximately 3 years; you will receive study medications for the duration of the study.

Anti-HIV drug regimens that include protease inhibitors (PIs) are very good at lowering viral load. However, some patients have a rise in HIV levels while on PI maintenance. It may be possible to keep HIV levels low using another class of drugs for maintenance that are easier to take and less expensive than PIs. If viral load increases while a patient is taking this second group of drugs, it may be possible to restart the PI drug regimen and again decrease HIV levels.

DETAILED DESCRIPTION:
Combination antiretroviral therapies using protease inhibitors (PIs) are capable of suppressing plasma HIV RNA to undetectable levels. However, approximately 10% of patients who achieve undetectable viral loads will experience a detectable rise in HIV RNA each year. When HIV replication has been suppressed to very low levels, it may be possible to consolidate antiretroviral therapy into a simpler and potentially less toxic "maintenance" regimen without a PI. Such a regimen would ideally be potent enough to continue to maintain viral suppression but use agents that are better tolerated, more easily salvaged, less expensive, and/or more convenient than PI-containing regimens. Subsequent rises in HIV viremia with non-PI maintenance regimens may respond to resumption of the pre-maintenance PI-containing regimen, extending the use of the potent PI class.

Patients are randomized 1:1:1 to treatment with ddI/d4T/HU (Arm A) versus ddI/d4T/EFV (Arm B) versus continuation of the pre-entry PI-containing regimen (Arm C). Viral load is measured at Weeks 1, 2, 4, 8, 12, 16, 20, and 24, then every 8 weeks for up to 3 years. Upon virologic failure (plasma HIV RNA greater than or equal to 200 copies/ml), or drug intolerance, patients on the maintenance regimens (Arms A and B) restart their pre-entry PI-containing regimen. Patients on Arm C are managed according to best medical judgment of their primary care provider in the event of virologic failure.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 13 years old (need consent if under 18).
* Are HIV-positive.
* Are taking your first anti-HIV drug regimen, which must include a PI and at least one NRTI (nucleoside reverse transcriptase inhibitor) and have been on this regimen for at least 12 months.
* Have a viral load less than 400 copies/ml for at least 12 months prior to study entry, and have a viral load less than 50 copies/ml within 60 days of study entry.
* Have a CD4 cell count of at least 200 cells/mm3 within 60 days of study entry.
* Are willing to go back on the drugs you are currently on, if necessary.
* Are willing to use effective methods of birth control during the study and for 3 months after.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken ddI, d4T, or HU for more than 2 weeks.
* Have taken any NNRTI (non-nucleoside reverse transcriptase inhibitor) for more than 7 days.
* Have ever taken EFV.
* Have received an HIV vaccine within 30 days prior to study entry.
* Have an AIDS-related cancer that requires chemotherapy.
* Have or have had pancreatic disease.
* Are being treated for a significant illness.
* Abuse drugs or alcohol.
* Are pregnant or breast-feeding.
* Are allergic to any study drugs.
* Have received certain medications.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wohl, Study Chair; Joe Eron, Study Chair; Roy Gulick, Study Chair
Locations (19):
- United States (19):
  - Willow Clinic, Menlo Park, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania